CLINICAL TRIAL: NCT01665859
Title: Nationwide Prospective Study of Surgical Risk Factors for Poor Outcome After Epigastric and Umbilical Hernia Repair
Brief Title: Risk Factors for Poor Outcome After Epigastric and Umbilical Hernia Repair
Status: Completed | Type: Observational
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Frederik Helgstrand, MD, Zealand University Hospital
Other Study IDs: FH09
Record Dates: First submitted 2012-08-13; First posted 2012-08-15 (Estimated); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Umbilical Hernia; Epigastric Hernia
Keywords: readmission; recurrence; umbilical; epigastric; hernia; outcome; morbidity
MeSH Terms: conditions — Hernia, Umbilical; Recurrence; Hernia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Danish Ventral Hernia Database: Patients registered in the Danish Ventral Hernia Database during January 1st 2007 to december 31st 2010

SUMMARY:
Umbilical and epigastric hernia repairs are common and performed by numerous surgical techniques. Considering that the hernia repairs in general are relatively small and simple procedures there are disproportionate poor results.

The aim of present study is to determine surgical risk factors for readmission after umbilical and epigastric hernia repair and to report risk factors for later reoperation for recurrence.

DETAILED DESCRIPTION:
All elective umbilical or epigastric hernias registered in the Danish Ventral Hernia Database are included in the study. The included patients will be followed in up to 4 years in order to identify correlation between technical aspects of the hernia repair and postoperative morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Umbilical or epigastric hernia repair

Exclusion Criteria:

-

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All elective umbilical or epigastric hernia repairs registered in tha Danish National Hernia Database from January 1st 2007 to December 31st 2010
Sampling Method: Non-Probability Sample
Enrollment: 6783 (Actual)
Dates: Start 2007-01; Primary Completion 2011-01 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
readmission | 30 days
  Riskfactors for readmission within 30 days after umbilical or epigastric hernia repair

SECONDARY OUTCOMES:
reoperation for recurrence | up to 4 years
  Risk factors for recurrence repair after umbilical or epigastric hernia repair

CONTACTS AND LOCATIONS:
Overall Officials: Frederik Helgstrand, MD, Principal Investigator — dept. surgery, Køge sygehus, Denmark
Locations (1):
- Køge Hospital, Køge, Denmark